CLINICAL TRIAL: NCT06444100
Title: Predictors of Child Abuse Among School Going Children and Impact of Structural Training on Child Abuse Among School Teachers of Dhulikhel Municipality
Brief Title: Predictors of Child Abuse Among School Going Children and the Impact of Structural Training on Child Abuse Among School Teachers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sita Karki, Associate Professor, Kathmandu University School of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35_2024
Record Dates: First submitted 2024-05-16; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Child Abuse

STUDY DESIGN:
Intervention Model Description: Selected schools will be divided into two groups: an intervention group, where teachers of selected schools will receive training on child abuse, and a control group without training. A comparative analysis will then evaluate the effectiveness of the intervention by assessing teachers' knowledge and attitudes towards child abuse. A pretest will be conducted to assess the existing knowledge level and attitude of the teachers toward child abuse. A 5-hour training session, led by an expert team, will follow the pretest questionnaire administration to all participants. The training will cover the introduction, definition, risk factors, signs, symptoms, and management of child abuse. Teachers will also be educated on how to report instances of child abuse.
  The training will incorporate interactive lectures, group discussions, and role-playing to effectively convey the management of child abuse. A post-test will be administered using the same questionnaires two weeks after the training
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will undergo training on child abuse led by an expert group, while the control arm will not receive this training. Both groups will undergo pre-testing before the intervention, followed by post-testing two weeks after the training period.
  Interventions: Procedure: Impact of structural training on child abuse
- Control (No Intervention): The control arm will not get any training.

INTERVENTIONS:
Procedure: Impact of structural training on child abuse — A focus group discussion to delve into teachers' perceptions of child abuse. Based on the findings, the training module will be modified as need-based.
  Phase II: Randomly selected samples will be invited, with the researcher explaining the study procedures and obtaining verbal and written consent from teachers and assent from children. A dedicated room will be arranged for data collection, and participants will be instructed on how to respond to child abuse questions on tablets.
  Phase-III A pretest will be conducted to assess the existing knowledge level and attitude of the teachers toward child abuse. A 5-hour training session, led by an expert team, will follow the pretest questionnaire administration to all participants. Teachers will also be educated on how to report instances of child abuse. A post-test will be administered using the same questionnaires two weeks after the training.
  Arms: Intervention

SUMMARY:
Child abuse stands as a global public health crisis, impeding the natural growth and development of children. The repercussions of abuse extend beyond immediate trauma, resulting in heightened medical costs and enduring health consequences that may persist into adulthood. These consequences encompass a spectrum of issues, including attachment disorders, behavioral abnormalities, depression, post-traumatic stress disorder, altered neurobiological structures, suicidal ideation, risky sexual practices, and susceptibility to sexually transmitted infections. The detrimental impact of any form of child abuse lingers into the adult lives of affected individuals.

This study aims to determine the Predictors of Child Abuse among School Going Children and the Impact of Structural Training on Child Abuse Among School Teachers of Dhulikhel Municipality in selected schools of Dhulikhel Municipality. Employing descriptive-analytical, true-experimental, and qualitative research designs, the study involves children aged ≥ 11 and teachers across diverse schools. A purposeful sample technique will be used to select teachers to explore school teachers' strategies in supporting students experiencing childhood violence. A simple stratified sampling technique will be used to select schools and a simple random sampling technique will be used to select the required number of students. Subsequently, one group of teachers undergoes comprehensive training on child protection recognition and response, while another does not. Following a two-week intervention, Investigators will conduct a posttest to evaluate teachers' knowledge and attitudes. To ensure clarity, both standard and self-constructed research tools will be translated into Nepali. Subsequently, these tools will be employed for data collection. The gathered information will be entered into an Excel datasheet and later transferred to Stata version 13 for a comprehensive analysis involving both descriptive and inferential statistics.

DETAILED DESCRIPTION:
This study aims to determine Predictors of Child Abuse among School Going Children and Impact of Structural Training on Child Abuse Among School Teachers of Dhulikhel Municipality in selected schools of Dhulikhel Municipality. Employing descriptive-analytical, true-experimental, and qualitative research designs, the study involves children aged ≥ 11 and teachers across diverse schools Study Population The participants-I Investigator purposefully selected teachers who are teaching in private and public schools of Dhulikhel municipality. The participants-II All children aged 11-18 years of age studying in different schools (public and private) of Dhulikhel Municipality. The participants-III Teachers are teaching in different schools in Dhulikhel Municipality which are selected by using a stratified random sampling technique.

Number of participants and Justification :

The first type of participants is 20-30 for focus group discussion. (3-5 group) The second type of participant is 421 students which is based on sample size calculation.

The Third type of participant is 206 teachers which is based on sample size calculation by taking 40% of the mean different knowledge score /SD to maintain optimum sample size.

Sampling Technique Sample-I Among the 26 schools, there are 8 private schools and 18 government schools. A stratified random sampling technique will be used to select 50% of the schools. From these selected schools, a list of teachers was obtained and categorized based on age, education level, gender, experience, and ethnic group. The required sample numbers will be purposefully selected from these groups, considering their characteristics such as interest and expressiveness. Sample-II In Dhulikhel Municipality, there are a total of 26 schools, encompassing both public and private institutions. To ensure a representative sample, 50% of these schools will be chosen utilizing the stratified random sampling technique. This method involves categorizing the schools based on certain criteria and then randomly selecting schools from each category. Subsequently, a proportionate stratified sampling technique will be employed to determine the necessary number of students from the selected schools. From these chosen schools, classes spanning grades 6 to 12 will be selected using a simple random sampling technique. To ensure a representative group, a proportionnâtes stratified sampling technique will be applied to determine the required number of participants. Sample-III Selected schools will be divided into two groups: an intervention group, where teachers of selected schools will receive training on child abuse, and a control group without training. A comparative analysis will then evaluate the effectiveness of the intervention by assessing teachers' knowledge and attitudes towards child abuse.

Criteria for sample selection Inclusion criteria: The teachers who are teaching in different schools of Dhulikhel Municipality. Exclusion criteria: The teachers who are not available during data collection are not interested and do not give consent to be involved as a participants. Inclusion criteria: The students who are aged 11-18 years old and willing to participate in the study. Exclusion criteria: The students who are sick, unable to understand the Nepali language, and do not give assent for participation in the study. Inclusion criteria: Teachers are teaching in different schools of Dhulikhel Municipality. Exclusion criteria: Teachers are unable to speak the Nepali language and unavailable during data collection.

Data Collection Technique Informed written consent will be obtained from participants after providing comprehensive study information. The study will utilize a focus group discussion to delve into teachers' perceptions of child abuse. The discussion will continue until data saturation is achieved. Randomly selected samples will be invited, with the researcher explaining the study procedures and obtaining both verbal and written consent from teachers, along with assent from children. A dedicated room will be arranged for data collection, and participants will be instructed on how to respond to questions on tablets. Any instances of child abuse identified during data collection will be promptly referred to the OCMC of Dhulikhel Hospital for further management as needed. Participants will receive a diary and pen after being informed about child abuse, as per the Protocol's instructions40. A pretest will be conducted to assess the existing knowledge level and attitude of the teachers toward child abuse. A 5-hour training session, led by an expert team, will follow the pretest questionnaire administration to all participants. The training will cover the introduction, definition, risk factors, signs, symptoms, and management of child abuse. Teachers will also be educated on how to report instances of child abuse. The training will incorporate interactive lectures, group discussions, and role-playing to effectively convey the management of child abuse. A post-test will be administered using the same questionnaires two weeks after the training.

Data collection tools The first part of the study is to assess school teachers' perceptions of child abuse. The focus group discussion will be done by using a self-constructed topic guide. The International Society for the Prevention of Abuse and Neglect (ISPCAN) and United Nations Children's Fund (UNICEF) have developed three questionnaires (one for parents, the ICAST-P; one for young adults, the ICAST-R; and one for children, the ICAST-C) to examine types of victimizations of childhood around the world. The researcher is going to use the ICAST-C tool to assess the prevalence of child abuse in Nepal.The prevalence of child abuse will be assessed using validated outcome measures like ICAST-C (ver3.0 children version) 41. Part-III Self constructed research tool tool will be used to assess knowledge and attitude of teachers toward child abuse.

Pretesting Moc test will be done before the finalization of the topic guide. Pre-testing the data collection tool: Pre-test will be performed on 10% of the total sample size in Banepa Municipality which will not be included in the main study. - Response and feedback will be taken and consulted with the research advisors.

Validity and reliability of tool The validated research tool will be translated into the Nepali language for its simplicity and comprehensibility. The pretest will be done in a 10% sample which will be excluded from the main study. Validity of the tool Content validity of the tool will be maintained by: -consulting with the research advisor, - subject expertise and concern authority, -review of the literature, and pretesting. Pre-testing the data collection tool: Pre-test will be performed on 10% of the total sample size in Banepa Municipality which will not be included in the main study. - Response and feedback will be taken and consulted with the research advisors.

Plan for supervision and monitoring In order to ensure the success and reliability of our research, a robust plan for supervision and monitoring during data collection is imperative. Investigators will begin by clearly defining the research objectives and establishing the guiding principles for our study. A detailed protocol will be crafted, covering every step from participant recruitment to data analysis. Thorough training sessions will be conducted to equip our team with the necessary skills, emphasizing the importance of consistency and accuracy. A well-defined supervision structure, led by a designated supervisor, will oversee the entire process. Regular check-ins, both scheduled and random, will be implemented to monitor progress, address challenges, and maintain alignment with research goals. Continuous data quality checks, a feedback mechanism, and comprehensive documentation will ensure the integrity of our data. Prior to full-scale data collection, a pilot test will be conducted to identify and address potential issues. Adherence to ethical standards, random spot checks, continuous training, and an emergency response plan will further fortify the robustness of our approach. This holistic plan aims to create a proactive and adaptive environment, ensuring the smooth execution of our research endeavors.

ELIGIBILITY:
Inclusion Criteria:

* Teachers from various selected secondary schools, both public and private, in Dhulikhel Municipality, Nepal.

Exclusion Criteria:

* Teachers from primary-level schools and refuse to take part in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Predictors of Child Abuse among School Going Children | 1 year
  Schools will be chosen through simple stratified sampling, and students via simple random sampling.The prevalence of child abuse will be assessed using the Child Abuse Screening Tool for Children (ICAST-C) through anonymous and ethically sound surveys.

SECONDARY OUTCOMES:
Impact of Structural Training on Child Abuse Among School Teachers in selected schools of Dhulikhel Municipality | 6 months
  Schools will be chosen through simple stratified sampling, and students via simple random sampling. One group of teachers will receive comprehensive training on child protection, while another will not. A pretest will assess teachers' existing knowledge and attitudes. Subsequently, all participants will undergo a 5-hour training session covering various aspects of recognizing and responding to child abuse followed by a post-test after a two-week training intervention to assess teachers' knowledge and attitudes towards child abuse.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandel P, Kunwar R, Karki S, Kandel D, Lamichhane P. Child maltreatment in Nepal: prevalence and associated factors. Public Health. 2017 Oct;151:106-113. doi: 10.1016/j.puhe.2017.06.020. Epub 2017 Jul 29. PMID 28763786
- [Background] Kumar MT, Kumar S, Singh SP, Kar N. Prevalence of child abuse in school environment in Kerala, India: An ICAST-CI based survey. Child Abuse Negl. 2017 Aug;70:356-363. doi: 10.1016/j.chiabu.2017.06.025. Epub 2017 Jul 7. PMID 28692832
- [Background] Kvist T, Dahllof G, Svedin CG, Annerback EM. Child physical abuse, declining trend in prevalence over 10 years in Sweden. Acta Paediatr. 2020 Jul;109(7):1400-1408. doi: 10.1111/apa.15215. Epub 2020 Mar 6. PMID 32031703
- [Background] Miragoli S, Balzarotti S, Camisasca E, Di Blasio P. Parents' perception of child behavior, parenting stress, and child abuse potential: Individual and partner influences. Child Abuse Negl. 2018 Oct;84:146-156. doi: 10.1016/j.chiabu.2018.07.034. Epub 2018 Aug 9. PMID 30099228
- [Background] Neupane D, Bhandari PM, Thapa K, Bhochhibhoya S, Rijal S, Pathak RP. Self-reported child abuse in the home: a cross-sectional survey of prevalence, perpetrator characteristics and correlates among public secondary school students in Kathmandu, Nepal. BMJ Open. 2018 Jun 19;8(6):e018922. doi: 10.1136/bmjopen-2017-018922. PMID 29921678
- [Background] Shrestha S, Baskota S, Karki U, Poudel L, Bhandari N, Gurung M, Rajbhandari B, Shrestha P. Child Sexual Abuse among School Children of a Municipality: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2021 Jul 30;59(239):672-677. doi: 10.31729/jnma.6865. PMID 34508495
- [Background] Song Y, Ji CY, Agardh A. Sexual coercion and health-risk behaviors among urban Chinese high school students. Glob Health Action. 2014 May 14;7:24418. doi: 10.3402/gha.v7.24418. eCollection 2014. PMID 24836445
- [Background] Tang CS. Childhood experience of sexual abuse among Hong Kong Chinese college students. Child Abuse Negl. 2002 Jan;26(1):23-37. doi: 10.1016/s0145-2134(01)00306-4. PMID 11860160